CLINICAL TRIAL: NCT01752153
Title: Immunomodulatory Effects of Silymarin in Patients With Beta-Thalassemia Major
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Marjan Gharagozloo, Assistant professor, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1929
Record Dates: First submitted 2012-11-21; First posted 2012-12-19 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-11

CONDITIONS: Immune Abnormalities
Keywords: Focus; immunomodulatory effect; of silymarin; on cell mediated immunity; Beta-Thalassemia; major patients.
MeSH Terms: conditions — beta-Thalassemia | interventions — Deferoxamine; Silymarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Silymarin (Legalon) (Experimental): Patients who were unable or unwilling to use desferrioxamine or had stopped desferrioxamine treatment for at least 6 months, were received only silymarin.
  Interventions: Drug: Silymarin (Legalon)
- Combined therapy (Deaferrioxamine+Silymarin (Legalon) (Experimental): In combined therapy group, patients continued desferrioxamine (Novartis Pharma AG, Switzerland) at the dose of 40 mg/Kg/day and Legalon® tablets (Madaus Pharma, Italy) was added to desferrioxamine regimen at the dose of 140 mg, taken orally, three times a day, 7 days a week.
  Interventions: Drug: Desferrioxamine, Legalon® (Silymarin)

INTERVENTIONS:
Drug: Desferrioxamine, Legalon® (Silymarin) — Desferrioxamine (Novartis Pharma AG, Switzerland) at the dose of 40 mg/Kg/day and Legalon® tablets (Madaus Pharma, Italy)
  Arms: Combined therapy (Deaferrioxamine+Silymarin (Legalon)
Drug: Silymarin (Legalon)
  Arms: Silymarin (Legalon)

SUMMARY:
A wide spectrum of immune abnormalities has been described by numerous studies involving β-thalassemic patients with multiple transfusions. The abnormalities observed are both quantitative and functional, and concern several components of the immune response. Flavonoids are phenolic compounds widely distributed in plants, which were reported to exert multiple biological effects, including antioxidant and free radical scavenging abilities. Silymarin, a flavonolignan complex isolated from milk thistle (Silybum marianum L. Gaertn), have been classified as cytoprotective, antioxidant, anti-inflammatory, and especially as hepatoprotective agents. Silymarin is already being used clinically for treatment of liver diseases.It is considered safe and well-tolerated, with reported adverse events similar to placebo. Several studies have also reported immunomodulatory actions of silymarin. It increases lymphocyte proliferation, interferon gamma, interleukin (IL)-4 and IL-10 secretions by stimulated lymphocytes in a dose-dependent manner. It has been shown that in vitro treatment of peripheral blood mononuclear cells with silymarin causes restoration of the thiol status and increases in T cell proliferation and activation. Because reactive oxygen species and iron overload play important roles in the pathophysiology of thalassemia, silymarin may be an effective therapy due to its antioxidant, immunomodulatory, cytoprotective and iron chelating activities. The present study designed to investigate the therapeutic activity of orally administered silymarin for treatment of β-thalassemia major, a well-known and prevalent disease in Iran, which is associated with oxidative stress, iron overload and immune abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Homozygous beta-thalassemia major
* Regularly blood transfusion
* Iron chelation therapy with subcutaneous desferrioxamine (DFO)40.0 mg/Kg/day for 5-7 days/week

Exclusion Criteria:

* Chronic hepatitis B infection
* Active hepatitis C infection
* A history of a positive HIV test
* Chronic renal or heart failure
* Iron chelation therapy with deferiprone
* Pregnancy
* Gastrointestinal conditions preventing absorption of an oral medication o
* noncompliance with prescribed therapy

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in T cell proliferation | 12 weeks
  PHA-activated T Cell Proliferation in Cell Culture was studied by Brdu Incorporation ELISA-based Assay
Changes from baseline the percentage of lymphocyte subsets | 12 weeks
  The percentage of T cell, B cell, and NK cells were studied using flowcytometry
Changes from baseline the production of cytokines in activated T cells | 12 weeks
  The concentrations of IL-2, IL-4, and IFN-gamma in supernatant of activated T cells were measured using ELISA assay.

CONTACTS AND LOCATIONS:
Overall Officials: Zahra Amirghofran, PhD, Study Director — Shiraz University of Medical Sciences
Locations (1):
- Department of Immunology, School of Medicine, Shiraz University of Medical Sciences, Shiraz, Fars, Iran